CLINICAL TRIAL: NCT00245297
Title: A Patient-Blinded, Randomized, Comparative, Multicenter, Crossover, (Liposome) Dose Finding Study of the Efficacy of Human Recombinant Factor VIII (Kogenate FS) Reconstituted in Pegylated Liposomes.
Brief Title: Study of the Efficacy of Human Recombinant Factor VIII (Kogenate FS) Reconstituted in Pegylated Liposomes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recoly N.V. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OMRI Lip-FVIII-05-1
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-10

CONDITIONS: Haemophilia A
Keywords: Bleeding disorder; severe Haemophilia A; Prophylaxis
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders | interventions — F8 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Kogenate FS, reconstituted in a suspension of liposomes

SUMMARY:
Primary efficacy endpoint: To study whether there is a difference in the length of the bleeding free periods between infusion of FVIII that is reconstituted with 22.1, 12.6, or 4.2 mg of pegylated liposomes per kg bwt compared with standard formulation.

Safety endpoint: To study the safety and tolerability of Kogenate FS reconstituted with Pegylated liposomes

DETAILED DESCRIPTION:
Each subject will receive treatment for three bleeding episodes ("wash-in", on demand injections) followed by a minimum 4 day wash-out. Following this each subject will be randomized to a specific treatment order. Each order consists of four identical blocks. In each block the following three injections will be given: 1 One prophylactic treatment (randomized solution for dissolution) 2 and 3. Two standard on-demand treatments for a spontaneous bleeding episode (standard Kogenate FS). Each block will be followed by a four day wash-out. In total each subject should receive 3+4x3=15 injections. It is estimated that each subject will be in the study for about 4 months. A treatment for a spontaneous bleeding episode may require more than one infusion.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age
* Severe haemophilia A (≤ 1% of baseline Factor VIII activity)
* At least 250 treatment cumulative exposure-days (CEDs) to previous products
* At least 25 cumulative exposure-days (CEDs) to previous products during one year prior to study start
* If HIV positive, CD4 lymphocytes ≥ 400/µl
* Subjects on demand treatment, and with a minimum bleeding/treatment pattern of a four episodes per month, evenly distributed within each month, during the three month preceding study start
* Subjects who have given their written informed consent.

Exclusion Criteria:

* Inhibitors or history of inhibitors
* History of adverse reactions related to Factor VIII
* Platelet count <90,000 /µl
* Subjects on prophylaxis treatment
* Subjects with concomitant debilitating disease (e.g. cancer, non-controlled diabetes, heart insufficiency, renal failure)
* Subjects with known sensitivity to blood products
* Subjects who have participated in another Ethical Committee approved Clinical Trial (including medical device studies) within the past 30 days
* Subjects with a weight over 86 kg or below 50 kg
* Subjects who do not understand or are not willing to comply with the requirement of the study protocol
* Subjects who cannot differentiate a bleeding episode from other causes of joint pain

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the number of bleeding free days (without a bleeding/treatment) between a randomized prophylactic infusion and following on demand injection. | Bleeding free time following four single doses will be studies

SECONDARY OUTCOMES:
In vivo recovery (IVR). | IVR will be performed at the first and last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Spira, MD. PhD., Study Director — Recoly C/o InSpira Medical AB, Nasbyv 38, 13553 Tyreso Sweden
Locations (3):
- Russia (3):
  - Center for Hematological Research, Department of Reconstructive Orthopedic Surgery, Moscow
  - The Russian Academy of Medical Sciences, Haemophilia Center, Moscow
  - Republic Haemophilia Center., Saint Petersburg

REFERENCES:
- [Background] Baru M, Carmel-Goren L, Barenholz Y, Dayan I, Ostropolets S, Slepoy I, Gvirtzer N, Fukson V, Spira J. Factor VIII efficient and specific non-covalent binding to PEGylated liposomes enables prolongation of its circulation time and haemostatic efficacy. Thromb Haemost. 2005 Jun;93(6):1061-8. doi: 10.1160/TH04-08-0485. PMID 15968389